CLINICAL TRIAL: NCT00002264
Title: Efficacy of Cow's Milk Immune Globulin in the Treatment of Chronic Intestinal Cryptosporidiosis in Patients With AIDS
Brief Title: The Effectiveness of Cow's Milk Immune Globulin in the Treatment of AIDS-Related Diarrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stolle Milk Biologic International (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 068A; WPC-S123
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-11

CONDITIONS: Cryptosporidiosis; HIV Infections
MeSH Terms: conditions — Cryptosporidiosis; HIV Infections

INTERVENTIONS:
Drug: Cryptosporidium Immune Whey Protein Concentrate (Bovine)

SUMMARY:
To examine the efficacy of cow's milk immune globulin in the treatment of diarrhea due to chronic intestinal cryptosporidiosis in patients with AIDS. The secondary end points of the study involve functional improvement which will be determined from nutritional and absorption studies.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Diagnosis of diarrhea associated with intestinal cryptosporidiosis.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Survival time projected to be < 9 weeks.
* Inability to tolerate any oral intake.
* Known allergy or intolerance to milk products.
* Organic mental syndrome precluding informed consent or following directions.

Patients with the following are excluded:

* Survival time projected to be < 9 weeks.
* Inability to tolerate any oral intake.
* Known allergy or intolerance to milk products.
* Organic mental syndrome precluding informed consent or following directions.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Luke's - Roosevelt Hosp Ctr, New York, New York, United States